CLINICAL TRIAL: NCT01230138
Title: A Randomised, Double Blind, Placebo Controlled Efficacy and Safety Trial of Different Doses/Dose Regimens of FP187 Compared to Placebo in Moderate to Severe Plaque Psoriasis (Pivotal Registration Study)
Brief Title: Pivotal Efficacy and Safety Registration Trial of FP187 in Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forward-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP187-201
Record Dates: First submitted 2010-09-24; First posted 2010-10-28 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- FP187 - TID (Experimental): FP187 250mg TID (total daily dose of 750mg)
  Interventions: Drug: FP187
- FP187- BID (Experimental): FP187 375mg BID (total daily dose of 750mg)of 750mg administered as 375mg BID
  Interventions: Drug: FP187
- FP187-LD-BID (Experimental): FP187 250mg BID (total daily dose of 500mg)
  Interventions: Drug: FP187
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo
- Open, flexible dosing treatment arm (Experimental): Open treatment using a flexible dosing schedule for 8 weeks with maximum dose of 750mg FP187 and with a total dosing of 20 weeks. All investigations following same schedule.
  Interventions: Drug: FP187

INTERVENTIONS:
Drug: Placebo — Placebo tablets
  Other Names: Placebo of FP187
  Arms: Placebo
Drug: FP187 — High daily dose of 750mg administered as 250mg TID
  Arms: FP187 - TID
Drug: FP187 — High daily dose of 750mg administered as 375mg BID
  Arms: FP187- BID
Drug: FP187 — Low daily dose of 500mg FP187 administered as 250mg BID
  Arms: FP187-LD-BID
Drug: FP187 — Oral tablets, up to 3 times daily for 20 weeks.
  Arms: Open, flexible dosing treatment arm

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of different doses and dose administrations of FP187 compared to a placebo treatment in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The trial tests two different dose levels and two different daily dosing schedules (twice daily (BID) and three times daily (TID))over 20 weeks of treatment. Key is effect as measured by achievement of a 75% reduction in PASI after 20 weeks and safety monitored by adverse events and safety lab.

There are 3 active arms:

1. FP-187 at a daily dose of 750mg divided in three doses (250mg TID)
2. FP-187 at a daily dose of 750mg divided in two doses (375mg BID)
3. FP-187 at a daily dose of 500mg divided in two doses (250mg BID)

and 1 placebo arm.

An additional open (flexible dosing) treatment arm has been amended to the trial

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex at least 18 years of age
* A clinical diagnosis of plaque psoriasis defined as skin areas with erythema, induration and scaling, with a body surface area of no less than 10% and in total to be scoring at least 10 on the PASI scale
* The psoriasis disease have been stable for at least 6 months at randomization
* Signed and dated informed consent
* Sexually active females of childbearing potential must be either surgically sterile (hysterectomy or tubal ligation) or use a highly effective (failure rate < 1%) medically accepted contraceptive method during the trial as well as one month after trial is finished such as:

  * Systemic contraceptive (oral, implant, injection),
  * Intrauterine device (IUD) inserted for at least one month prior to study entrance
* Willingness and ability to comply with the trial procedures
* Patient is beside the psoriasis disease in good general health in the opinion of the Investigator, as determined by medical history, physical examination, vital signs and clinical laboratory parameters (hematology, biochemistry and urinalysis).

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding or planning to become pregnant up to 7 months from treatment start as well as male patients plan-ning pregnancy with their partner up to 7 months from treatment start or practise unprotected sexual relationship up to 7 months from treatment start
* Known allergy to any of the constituents of the product being tested
* Pustular forms of psoriasis, erythrodermic or guttate psoriasis
* Known immunosuppressive diseases (e.g., AIDS/HIV)
* Presence of another serious or progressive disease which, according to the Investigator may interfere with treatment outcome
* Active skin disease such as atopic dermatitis, rosacea, lupus erythematosus, or other inflammatory or infectious skin disease which, according to the Investigator may interfere with treatment outcome
* Use of topical medical treatment or UVB treatment - Use of systemic anti-psoriatic treatment preceding the baseline visit Methotrexate, cyclosporine, steroids or PUVA treatment within x weeks; Biological treatment (efalizumab, adalimumab, infliximab, etanercept) within xx weeks; Acitretin within x months; Treatment with Fumaderm® or other DMF containing products during past xx weeks prior to baseline visit; Discontinuation of previous treatment with Fumaderm® or other DMF containing products due to lack of efficacy or side effects;
* Has within the past x weeks prior to baseline visit been treated with drugs influencing the course of the psoriasis such as antimalarial drugs, beta-blockers or lithium
* Has a relevant clinical history of stomach or intestinal problems (eg gastritis or peptic ulcer within the last 10 years )
* Has liver enzyme measures (AST, ALT, Gamma-GT) higher than 2x UNL)
* Has an estimated Creatinine Clearance: < xx ml/min
* Has leucopenia (leukocyte count < x/mm3) or eosinophilia (count >x/µl) or lymphopenia (count < x/nl).
* Has protein in the urine test at screening or baseline visit
* Participation in another clinical trial during the last month preceding the baseline visit or participation in a trial with treatment of biologicals within x months prior to baseline visit
* Patients who are involved in the organisation of the clinical investigation or are in any way dependant on the investigator or sponsor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving PASI 75 compared to placebo | After 20 weeks of treatment
  Proportion of patients achieving PASI75 (a reduction in the PASI score of 75% or more)

SECONDARY OUTCOMES:
PASI 75 | At week 4, 8, 12 and 16
  Proportion of patients achieving PASI75 (a reduction of the PASI score of 75% or more compared to baseline)
PASI 50 | At week 4, 8, 12, 16 and 20
  Proportion of patients who achieves PASI 50 (a reduction of the PASI score of 50% or more compared to baseline)
PASI 90 | At week 4, 8, 12, 16 and 20
  Proportion of patients achieving PASI90 (a reduction of the PASI score of 90% or more compared to baseline
PGA (Physicians Global Assessment) | At week 4, 8, 12, 16 and 20
  On a 5-point scale from 0 (abscence or very mild disease) to 4 (very severe disease) proportion of patients being responders - defined as patients achieving either a score of 0 or 1 or a two point improvement
PaGA (Patients Global Assessment | At week 4,8,12,16 and 20
  Patients evaluation on a 5-point Likert scale 1 (very good) - 5 (very poor)based on the evaluation of: "Considering all the ways your psoriasis affects you, how have you been doing in the last 24 hours?"
Pruritus | At week 4, 8, 12, 16 and 20
  Patient evaluation of pruritus measured on a VAS (Visual Analog Scale) from 0mm (no pruritus) to 100mm (worst possible pruritus)
Patient rated QoL (Quality of Life) | At week 4, 8, 12, 16 and 20
  Patient filling in 10 questions on the DLQI QoL system with a calculated summary score and analysis of the improvement from baseline
Adverse events (AEs) | At week 4, 8, 12, 16 and 20
  Summary of incidense and severity of AEs and ADRs (Adverse Drug Reactions)/SAEs (Serious Adverse Events)/SUSARs (Suspected Unexpected Serious Adverse Reactions)
Safety lab test | At week 20
  Summary of lab parameters and clinically relevant changes over the treatment period in standard clinical chemistry tests, standard haematology tests and urin dip stick test

CONTACTS AND LOCATIONS:
Overall Officials: Peder M Andersen, MD, Study Director — Forward-Pharma GmbH
Locations (2):
- Germany (2):
  - Dermatological Dept., Uniklinikum, TU-Dresden, Dresden
  - SCIderm, Hamburg

REFERENCES:
- See also: Web page of Forward Pharma — http://www.forward-pharma.com